CLINICAL TRIAL: NCT01372462
Title: A Pilot Study of the Physiologic Effects of Using the Breathe Technologies Noninvasive Open Ventilation System During Constant Work Rate Exercise in Subjects With Chronic Obstructive Pulmonary Disease
Brief Title: Effects of the Breathe Technologies Ventilation System in Subjects With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Breathe Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CP-00-0035
Record Dates: First submitted 2011-06-07; First posted 2011-06-14 (Estimated); Results first posted 2016-10-12 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Ventilator; Constant work rate
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Cannula

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- NIOV - Room air (Experimental): Subjects exercise using the NIOV device powered by compressed air (room air, 21% O2).
  Interventions: Device: NIOV - Room Air
- NIOV - Oxygen (Experimental): Subjects exercise using the NIOV device powered by compressed medical oxygen (100% O2).
  Interventions: Device: NIOV - Oxygen
- Nasal Cannula Oxygen (Active Comparator): Subjects exercise using a standard nasal cannula using medical oxygen (100% O2).
  Interventions: Device: Nasal Cannula Oxygen
- No treatment (No Intervention): Control arm. Subjects exercise without using supplemental oxygen or NIOV.

INTERVENTIONS:
Device: NIOV - Room Air — Noninvasive ventilation with device powered by compressed room air.
  Other Names: NIOV
  Arms: NIOV - Room air
Device: NIOV - Oxygen — Noninvasive ventilation with device powered by compressed medical (100%) oxygen.
  Other Names: NIOV
  Arms: NIOV - Oxygen
Device: Nasal Cannula Oxygen — Supplemental oxygen delivered using a standard nasal cannula connected to 100% medical oxygen.
  Other Names: Cannula
  Arms: Nasal Cannula Oxygen

SUMMARY:
Pilot study in 15 stable male subjects with severe-to-very severe Chronic Obstructive Pulmonary Disease (COPD) to evaluate the effects of short term use of the Breathe Technologies noninvasive open ventilation (NIOV) system on respiratory mechanics during constant work rate exercise in subjects with severe COPD.

DETAILED DESCRIPTION:
Study was a randomized double-blinded crossover design in which subjects completed a series of exercises at a constant work rate while using 1) Test noninvasive ventilation (NIOV) system powered by compressed air, 2) Test NIOV system powered by 100% oxygen, 3) nasal cannula oxygen, 4) nothing (Control). Subjects were assessed during constant work rate exercise as reflected by exercise duration, isotime oxygenation (SpO2), and isotime dyspnea score (Borg). Exercise sessions took place over 4 visits with each visit lasting approximately 5 hours.

ELIGIBILITY:
Inclusion Criteria:

* Adult males, ≥ 40 years of age
* Diagnosis of severe COPD (GOLD stage III or IV) defined as having a FEV1 < 50% of predicted and an FEV1/FVC ratio < 70% of predicted
* Ventilatory limitation to exercise, documented by a VE/MVV > 0.85
* SpO2 between 80% and 88% during incremental exercise testing on room air
* Willingness and ability (after training) to exercise on a cycle ergometer
* Willingness and ability to perform all other study related procedures and tasks
* Ability to be properly fitted with the Breathe nasal mask
* Ability to tolerate and be appropriately titrated on the Breathe ventilator (See Appendix E)
* Ability to be properly fitted with an exercise mask
* Fluency in written and spoken English
* Provision of written informed consent

Exclusion Criteria:

* History of acute exacerbation of COPD within 30 days of screening
* History of serious epistaxis within 14 days of screening
* Requirement of > 5 LPM nasal O2 to maintain an SpO2 > 90% while at rest
* History of pneumothorax secondary to lung bullae
* History of intolerance to supplemental oxygen
* Musculoskeletal or other non-pulmonary impairment that limits exercise tolerance
* Inability to achieve an optimal CWR level (4-7 minutes) during Study Visit 1R
* Current participation in another interventional study or participation within 14 days of screening
* Presence of any condition or abnormality that in the opinion of the Principal Investigator may compromise the subject's safety or the quality of the study data

Min Age: 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Casaburi, Ph.D., M.D., Principal Investigator — Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Locations (1):
- Harbor-UCLA Medical Center, Torrance, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: All subjects completed all 4 visit days in which they were randomized to receive which treatment to receive first: 1) NIOV - Oxygen, 2) NIOV - Room Air, 3) Oxygen Nasal Cannula, 4) No treatment.
  Study days 1,2,3, and 4; Day 1 for no treatment; day 2 for no treatment and NIOV - Room Air and NIOV - oxygen; Day 3 for no treatment and NIOV - Room Air and NIOV - oxygen; Day 4 for NIOV - oxygen and Nasal Cannula Oxygen.
Period: NIOV - Room Air
Arm/Group | All Study Participants
Started | 15
Completed | 15
Not Completed | 0
Period: NIOV - Oxygen
Arm/Group | All Study Participants
Started | 15
Completed | 15
Not Completed | 0
Period: Oxygen Nasal Cannula
Arm/Group | All Study Participants
Started | 15
Completed | 15
Not Completed | 0
Period: No Treatment Control
Arm/Group | All Study Participants
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The primary endpoint is difference in endurance between cannula oxygen and NIOV+O2. Assuming 153 sec clinically important difference, 183 sec SD of increase and α=0.05, a sample size of 15 yields 85% power.
Groups:
- Overall Study Group: Crossover design. Subject were randomized to complete all 4 study arms: 1) NIOV - Oxygen, 2) NIOV - Room Air, 3) Oxygen Nasal Cannula, 4) No treatment
Arm/Group | Overall Study Group
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Only male subjects were recruited due to need for placement of sensors on an exposed chest area.
  Participants
    Female | 0
    Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Exercise Duration for Constant Work Rate Exercise Tests Under 4 Test Conditions
Description: Mean differences between NIOV - oxygen, NIOV - Room Air, Nasal Cannula Oxygen, and no treatment (control).
Time Frame: Study days 1,2,3, and 4; Day 1 for no treatment; day 2 for no treatment and NIOV - Room Air and NIOV - oxygen; Day 3 for no treatment and NIOV - Room Air and NIOV - oxygen; Day 4 for NIOV - oxygen and Nasal Cannula Oxygen.
Population: Per protocol analysis
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | NIOV - Room Air | NIOV - Oxygen | Nasal Cannula Oxygen | No Treatment
Number analyzed (Participants) | 15 | 15 | 15 | 15
minutes | 6.3 (4.1) | 17.5 (5.7) | 11.4 (6.8) | 5.6 (1.9)
Statistical Analysis 1: Comparison: NIOV - Oxygen vs Nasal Cannula Oxygen; The primary endpoint was difference in endurance between nasal cannula oxygen and NIOV+O2. Assuming 153 sec clinically important difference, 183 sec SD, and α=0.05, a sample size of 15 yielded 85% power; Test type: Superiority or Other; p < 0.05, ANOVA; Newman-Keuls multiple comparisons test
Statistical Analysis 2: Comparison: NIOV - Room Air vs NIOV - Oxygen; Test type: Superiority or Other; p < 0.05, ANOVA
Statistical Analysis 3: Comparison: NIOV - Oxygen vs No Treatment; Test type: Superiority or Other; p < 0.05, ANOVA

2. Secondary Outcome: SpO2 During Constant Workrate Exercise at Isotime
Description: Mean differences between NIOV - oxygen, NIOV - Room Air, Nasal Cannula Oxygen, and no treatment (control).
Time Frame: Outcome was measured in each of the Study day 1,2, 3 and 4. Study days 1,2,3, and 4; Day 1 for no treatment; day 2 for no treatment and NIOV - Room Air and NIOV - oxygen; Day 3 for no treatment and NIOV - Room Air and NIOV - oxygen; Day 4 for NIOV - oxyg
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: percentage of oxyHb saturation
Arm/Group | NIOV - Room Air | NIOV - Oxygen | Nasal Cannula Oxygen | No Treatment
Number analyzed (Participants) | 15 | 15 | 15 | 15
percentage of oxyHb saturation | 87.9 (3.8) | 98.5 (1.0) | 92.7 (3.9) | 88.2 (2.2)
Statistical Analysis 1: Comparison: NIOV - Oxygen vs Nasal Cannula Oxygen; One-way, repeated-measures ANOVA and Newman-Keuls multiple comparisons test; Test type: Superiority or Other; p < 0.05, ANOVA; Newman-Keuls multiple comparisons test
Statistical Analysis 2: Comparison: NIOV - Room Air vs NIOV - Oxygen; Test type: Superiority or Other; p < 0.05, ANOVA
Statistical Analysis 3: Comparison: NIOV - Oxygen vs No Treatment; Test type: Superiority or Other; p < 0.05, ANOVA

3. Secondary Outcome: Borg Dyspnea Score During Constant Workrate Exercise at Isotime
Description: Mean differences between NIOV - oxygen, NIOV - Room Air, Nasal Cannula Oxygen, and no treatment (control) at isotime. Borg Dyspnea Score ranges in values from 0 to 10. The lower score represent better outcome.
  0 = No breathlessness at all, representing better outcome 10 = Maximum breathlessness, representing worse outcome
Time Frame: Outcome was measured in each Study day 1,2,3 and 4. Study days 1,2,3, and 4; Day 1 for no treatment; day 2 for no treatment and NIOV - Room Air and NIOV - oxygen; Day 3 for no treatment and NIOV - Room Air and NIOV - oxygen; Day 4 for NIOV - oxygen and N
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NIOV - Room Air | NIOV - Oxygen | Nasal Cannula Oxygen | No Treatment
Number analyzed (Participants) | 15 | 15 | 15 | 15
units on a scale | 3.3 (1.8) | 1.8 (1.3) | 2.5 (1.7) | 4.6 (2.0)
Statistical Analysis 1: Comparison: NIOV - Oxygen vs Nasal Cannula Oxygen; Per protocol; Test type: Superiority or Other; p < 0.05, ANOVA — One-way, repeated-measures ANOVA and Newman-Keuls multiple comparisons tests; Newman-Keuls multiple comparisons tests
Statistical Analysis 2: Comparison: NIOV - Room Air vs NIOV - Oxygen; Test type: Superiority or Other; p < 0.05, ANOVA
Statistical Analysis 3: Comparison: NIOV - Oxygen vs No Treatment; Test type: Superiority or Other; p < 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: Continuously for up to 8 hours on study days in which exercise testing was conducted
Arm/Group | NIOV - Room Air | NIOV - Oxygen | Nasal Cannula Oxygen | No Treatment
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No